CLINICAL TRIAL: NCT02551471
Title: Benchmarking Trial Between France and Australia Comparing Management of Primary Rectal Cancer Beyond TME (Total Mesorectum Excision) and Locally Recurrent Rectal Cancer
Acronym: PELVICARE
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2014/37
Record Dates: First submitted 2015-08-31; First posted 2015-09-16 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Rectal Cancer
Keywords: Locally advanced rectal cancer; Fixed primary rectal cancer; Pelvic recurrence; Benchmarking France Australia
MeSH Terms: conditions — Rectal Neoplasms | interventions — Magnetic Resonance Spectroscopy; Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- French patients
  Interventions: Other: Blinded inter-country reading of pelvic MRI (Magnetic Resonance Imaging); Other: MDT (Multidisciplinary team) meeting observation; Other: Semi-structured exploratory interviews and focus group with MDT health professional attendees
- Australians patients
  Interventions: Other: Blinded inter-country reading of pelvic MRI (Magnetic Resonance Imaging); Other: MDT (Multidisciplinary team) meeting observation; Other: Semi-structured exploratory interviews and focus group with MDT health professional attendees

INTERVENTIONS:
Other: Blinded inter-country reading of pelvic MRI (Magnetic Resonance Imaging) — This experiment will consist of an inter-country reading of patients' pelvic MRIs, "blind" to the other country's decision. The MRI shared will be the one based on which the treatment decision will be made. In case of medical contraindication to perform pelvic MRI, the scan will be used to assess the care-decision concordance between both countries.
Other: MDT (Multidisciplinary team) meeting observation — 3 per centre with "real" patient cases and "theoretical" patient cases (blinded pelvic MRI re-reading).
Other: Semi-structured exploratory interviews and focus group with MDT health professional attendees — Will identify care management systems for PRC-bTME and LRRC patients, explore social representations that direct the formulation of a therapeutic decisions and identify cultural, medical and personal factors

SUMMARY:
The incidence of rectal cancers is at 15,000 new cases per year in France of which 10 to 15% are locally advanced (T4bNxM0) at the moment of diagnosis. The rate of invaded resection margins (R1) for these locally advanced and fixed rectal tumours varies from 10 to 20%. The invasion of the resection margins triples the risk of local recurrence. In the absence of surgical treatment, the 5-year survival rate for patients having had pelvic recurrence of rectal cancer is lower than 4% whereas it varies from 35 to 40% in cases of curative resection. The care and management of locally advanced and fixed rectal tumours and pelvic recurrence of rectal cancer constitutes, therefore, in the absence of recommendation, a difficult therapeutic problem with great variability in the methods of care and management around the world. These variations in practice can be explained by structural and organizational differences, as well as cultural dissimilarities. With regards to the organization of its healthcare system, Australia is shown to be a leader as regards the care and management of locally advanced and fixed rectal tumours and pelvic recurrence of rectal cancer.

DETAILED DESCRIPTION:
This research project rests on the comparison between two contrasting countries with regards to the care management of PRC-bTME (Primary rectal cancer beyond total mesorectum excision planes) and LRRC (Locally recurrent rectal cancer), France and Australia. Regarding its healthcare system for patients with PRC-bTME and LRRC, Australia equipped itself with a veritable policy of centralisation and clinical pathway, appearing as an international referent country in this surgical field.

The main hypotheses of research are that these differences rest on individual and collective representation of disease, organisations, structures, clinical pathway and care management.

Benchmarking of clinical practices is a process that consists of a structured comparison and the sharing of good practices of clinical care; it is based on a quality of care assessment and allows to fit into an approach of continuous improvement of this quality of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients operable and/or capable of receiving a radiotherapy and/or a chemotherapy
* Patients in care in the French and Australian centres participating in the study

Exclusion Criteria:

* Patients suffering from primitive rectal cancer at a stage inferior to T4b
* Patients suffering from primitive locally-advanced metastatic rectal cancer (T4NxM1)
* Patients suffering from recurrence of metastatic rectal cancer
* Patients having been refused a surgical procedure because of one or multiple comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from primitive locally-advanced non-metastatic rectal cancer (T4bNxM0), operated and non-operated.
  Patients suffering from non-metastatic recurrence of rectal cancer, operated and non-operated
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Clinical resection rates in both countries | 12 months
  Expressed as a percentage and corresponding to the ratio between the number of patients operated and the number of patients discussed in colorectal MDT meetings for PRC-bTME and LRRC. These rates will be expressed separately in each country and compared.

SECONDARY OUTCOMES:
Concordance rate of operative decisions between France and Australia | 6 months, 12 months
  An analysis of concordance between French and Australian operative decisions will be carried out through the radiological (or theoretical) resectability rate, expressed as a percentage and corresponding, after blind inter-country reading of pelvic MRIs, to the ratio between the number of patients judged to have resectable tumours and the number of all MRI re-reading.
R0 resection rate | 12 months
  Expressed as a percentage and corresponding to the report of the number of patients operated with a surgical resection margin > 1mm on the number of operated patients
Disease Free Survival | 12 months
Overall Survival | 12 months
Post-operative morbidity and mortality rates | 30 days
  Evaluated according to the Dindo scale for patients in curative intent treatment. Grade I was any deviation from the normal postoperative course, Grade II included pharmacological treatment, Grade III was complications requiring surgical, endoscopic or radiological intervention, Grade IV included life-threatening complications requiring intensive care unit management and Grade V complications caused postoperative death.
Quality of life questionnaire | 6 months, 12 months
  According to MOS SF-36 score and FACT-C score
Stress level score | 6 months, 12 months
  According to distress thermometer (score range from 0 [no distress] to 10 [extreme distress])
Analyses of semi-structured interviews | 12 months
  Occurrence and cooccurrence computation of thematic contents (frequency and Chi square analyses) ; similarity analyses (maximum three with connectedness and similarity index computations, identification of the central and peripheral representation cores in each occupational group)

CONTACTS AND LOCATIONS:
Locations (12):
- Australia (2):
  - Peter Maccallum Cancer centre, Melbourne
  - Royal Prince Alfred Hospital Sydney, Sydney
- France (10):
  - Hôpital Saint-André, Bordeaux
  - Hopital Beaujon, Clichy
  - Hopital A.Michallon, Grenoble
  - Centre Oscar Lambret CLCC, Lille
  - Hopital Lyon Sud, Lyon
  - Institut Paoli Calmette, Marseille
  - CLCC Val d'Aurelle, Montpellier
  - Hôpital Saint-Antoine, Paris
  - Hopital Charles Nicolle, Rouen
  - Hôpital Purpan, Toulouse

REFERENCES:
- [Derived] Denost Q, Saillour F, Masya L, Martinaud HM, Guillon S, Kret M, Rullier E, Quintard B, Solomon M. Benchmarking trial between France and Australia comparing management of primary rectal cancer beyond TME and locally recurrent rectal cancer (PelviCare Trial): rationale and design. BMC Cancer. 2016 Apr 4;16:262. doi: 10.1186/s12885-016-2286-1. PMID 27044252